CLINICAL TRIAL: NCT01595282
Title: Intramuscular Ketorolac Versus Oral Ibuprofen for Pain Relief in First Trimester Suction Curettage: a Randomized Clinical Trial.
Brief Title: Intramuscular Ketorolac Versus Oral Ibuprofen for Pain Relief in First Trimester Suction Curettage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-p-000259
Record Dates: First submitted 2011-05-19; First posted 2012-05-10 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: pain; suction curettage
MeSH Terms: conditions — Pain | interventions — Ketorolac; Ketorolac Tromethamine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac (Experimental): Intramuscular injection of ketorolac 60 mg in 2cc -plus- placebo tablet (calcium carbonate 600 mg tablet). For subjects who are 50 kg or less, intramuscular injection of ketorolac 30 mg in 1cc -plus- placebo tablet (calcium carbonate 600 mg tablet)
  Interventions: Drug: Ketorolac
- Ibuprofen (Active Comparator): Ibuprofen 800 mg tablet -plus- intramuscular injection of 2cc saline placebo. For subjects weighing 50 kg or less, ibuprofen 600 mg tablet -plus- intramuscular injection of 2cc saline placebo
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ketorolac — For subjects weighing over 50 kg, ketorolac 60 mg in 2cc administered via intramuscular injection 30-60 minutes before suction curettage procedure. For subjects weighing 50 kg or less, ketorolac 30 mg in 1 cc administered via intramuscular injection 30-60 minutes before suction curettage procedure
  Other Names: Toradol
  Arms: Ketorolac
Drug: Ibuprofen — For subjects weighing over 50 kg, ibuprofen 800 mg tablet administered orally 60-90 minutes before suction curettage procedure. For subjects weighing 50 kg or less, ibuprofen 600 mg tablet administered orally 60-90 minutes before suction curettage procedure.
  Arms: Ibuprofen

SUMMARY:
The aim of this study is to compare the effect of pre-procedural ketorolac to ibuprofen on immediate post-procedural pain scores in patients undergoing first trimester suction curettage with local anesthesia only.

Our primary hypothesis is that IM ketorolac compared to oral ibuprofen will result in an approximate 30% reduction in pain scores on a 21-point numerical rating scale immediately after the procedure.

Secondary hypotheses include:

* Pain scores on the 21-point scale will also be significantly lower in the ketorolac group immediately after cervical dilation and 15 minutes post-procedure.
* Fewer patients in the ketorolac group will rate their pain as "severe" on a subjective pain rating scale.
* Patients in the ketorolac group will be more satisfied with their pain control.
* Side effects will be similar between groups.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 or older seeking suction curettage at Planned Parenthood League of Massachusetts (PPLM)
* Gestational age less than or equal to 11+6, confirmed by ultrasound
* Eligible for suction curettage according to PPLM protocols
* Choice of local anesthesia

Exclusion Criteria:

* Choice of IV sedation for pain control
* Hypersensitivity to NSAIDs or lidocaine
* Contraindications to NSAIDs:

Active renal disease Active hepatic disease Gastric ulcer disease or gastritis Long-term NSAID or aspirin use Bleeding disorder

* NSAIDs taken < 8 hours prior to procedure
* Need for cervical ripening with either misoprostol or mechanical priming agent (laminaria/Dilapan)
* Long-term narcotic use
* Unable or unwilling to complete required study procedures
* Previous participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, MPH, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: June 2011-May 2012
  Clinic: free-standing, outpatient health center
Period: Overall Study
Arm/Group | Ketorolac | Ibuprofen
Started | 47 | 47
Completed | 47 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Ibuprofen | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (6.4) | 25.3 (4.7) | 25.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 94
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African American/Black | 20 | 17 | 37
  White | 11 | 14 | 25
  Asian | 3 | 4 | 7
  Multiracial | 2 | 3 | 5
  Other | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Immediate Post-procedure Pain Score
Description: The primary endpoint is subjects' immediate post-procedure pain score on a 21-point 0 to 100 scale, 0 = no pain and 100 = worst possible pain (in increments of five). This scale has been previously validated and used for research purposes, including for pain research evaluating suction curettage elsewhere and at our institution (Jensen 1986, Williamson 2004, Allen 2009).
Time Frame: Immediately (within 1 minute) after suction and speculum removal
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ibuprofen
Number analyzed (Participants) | 47 | 47
units on a scale | 52.3 (29.1) | 56.2 (30.2)

2. Secondary Outcome: Pain Scores Immediately After Cervical Dilation
Description: 21-point 0 to 100 scale where 0 = no pain and 100 = worst possible pain (in increments of five)
Time Frame: Immediately (within 1 minute) after cervical dilation prior to the introduction of the suction cannula
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ibuprofen
Number analyzed (Participants) | 47 | 47
units on a scale | 41.6 (27.72) | 45.4 (28.54)

3. Secondary Outcome: Pain Scores 15 Minutes Post-procedure
Description: 21-point 0 to 100 scale, where 0 = no pain and 100 = worst possible pain (in increments of five)
Time Frame: Fifteen minutes after the procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Ibuprofen
Number analyzed (Participants) | 47 | 47
units on a scale | 22.3 (20.8) | 15.0 (17.3)

ADVERSE EVENTS:
Arm/Group | Ketorolac | Ibuprofen
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No